CLINICAL TRIAL: NCT00036348
Title: Study of Aripiprazole in Patients With a History of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-010
Record Dates: First submitted 2002-05-08; First posted 2002-05-10 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is effective in the treatment of patients with a history of bipolar disorder.

ELIGIBILITY:
Patients with a history of Bipolar I Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Tuscaloosa, Alabama
  - Local Institution, Chillicothe, California
  - Local Institution, Riverside, California
  - Local Institution, Stanford, California
  - Local Institution, Torrance, California
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Louisville, Kentucky
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Belmont, Massachusetts
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, New York, New York
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Memphis, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, San Antonio, Texas

REFERENCES:
- [Derived] Kemp DE, Calabrese JR, Tran QV, Pikalov A, Eudicone JM, Baker RA. Metabolic syndrome in patients enrolled in a clinical trial of aripiprazole in the maintenance treatment of bipolar I disorder: a post hoc analysis of a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2010 Sep;71(9):1138-44. doi: 10.4088/JCP.09m05159gre. Epub 2010 May 4. PMID 20492838
- [Derived] Muzina DJ, Momah C, Eudicone JM, Pikalov A, McQuade RD, Marcus RN, Sanchez R, Carlson BX. Aripiprazole monotherapy in patients with rapid-cycling bipolar I disorder: an analysis from a long-term, double-blind, placebo-controlled study. Int J Clin Pract. 2008 May;62(5):679-87. doi: 10.1111/j.1742-1241.2008.01735.x. Epub 2008 Mar 25. PMID 18373615
- [Derived] Keck PE Jr, Calabrese JR, McIntyre RS, McQuade RD, Carson WH, Eudicone JM, Carlson BX, Marcus RN, Sanchez R; Aripiprazole Study Group. Aripiprazole monotherapy for maintenance therapy in bipolar I disorder: a 100-week, double-blind study versus placebo. J Clin Psychiatry. 2007 Oct;68(10):1480-91. doi: 10.4088/jcp.v68n1003. PMID 17960961